CLINICAL TRIAL: NCT03629626
Title: A Prospective, Randomized Trial Comparing ERAS and Conventional Protocol for Perioperative Care of Patients After Gynecological Surgery
Brief Title: Enhanced Recovery After Surgery (ERAS) in Gynecological Surgery (ERASGS-01)
Acronym: ERAS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shandong University (Other)
Responsible Party: Principal Investigator, Beihua Kong, Clinical Professor, Shandong University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ERASGS-01
Record Dates: First submitted 2018-08-10; First posted 2018-08-14 (Actual); Last update posted 2023-04-25 (Actual); Status verified 2023-04

CONDITIONS: Gynecologic Disease; Gynecologic Cancer
Keywords: preoperative / intraoperative/ postoperative management
MeSH Terms: conditions — Genital Diseases, Female

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conventional Perioperative (SP) care (No Intervention): Conventional Perioperative (SP) care
- ERAS protocol (Experimental): preoperative / intraoperative/ postoperative management
  Interventions: Procedure: ERAS protocol

INTERVENTIONS:
Procedure: ERAS protocol — preoperative management Optimization of relevant medical uncontrolled situations, avoid fasting, avoid bowel preparation, avoid premedications, nutritional assessment, stop smoking, stop alcohol and appropriate counselling
  intraoperative management Multimodal prevention of prophylaxis against nausea and vomiting (PONV) (according to preoperative assessment of Apfel Score) with a combination of multiple antiemetic drugs.
  postoperative management Postoperative pain control is obtained with opioid sparing strategies, in order to avoid Post Operative Ileus (POI) and PONV.
  It is proposed to chew gum three times daily , fluid therapy, early mobilization, early feeding within 2 hours postoperative for at least 15 minutes and eventually to promote a faster bowel function.
  Arms: ERAS protocol

SUMMARY:
Enhanced recovery programs are composed of preoperative, intraoperative and postoperative strategies combined to form a multi-modal pathway. ERAS requires a multidisciplinary team of anesthetists, surgeons and nurses for successful implementation and realization of its advantages.The aim of this study is to compare outcomes of conventional perioperative care with those of an enhanced recovery after surgery (ERAS) perioperative care plan in women undergoing surgery for gynecologic cancer or suspected gynecologic disease.

DETAILED DESCRIPTION:
The study design is a two-arm, randomized, controlled trial. The control arm will consist of standard conventional perioperative care. The intervention arm will consist of a protocol-driven ERAS program. The investigators believe that this information will be very useful because although there is a national interest in creating ERAS protocols for gynecology, there currently is very little published on the subject. Investigators hypothesize that those patients randomized to the ERAS protocol will have shorter lengths of hospital stay and complications, without increasing readmission rates. The investigators would like to publish the investigators' results and protocol as a resource for other institutions to adopt.

ELIGIBILITY:
Inclusion Criteria:

* Age >18 and <70 years old
* Patients candidated for elective gynecological surgery for benign pathology
* Patients with diagnosis of gynecological neoplasm and candidated for elective gynecological surgery
* Signed consent form

Exclusion Criteria:

* Contraindication to loco-regional anaesthesia
* Patients with ileus or subocclusive condition prior surgery
* Coagulation disorders
* Organ failure or severe disfunction (heart, renal, pulmonary, hepatic)
* Uncontrolled hypertension (>180/95)
* Alcohol or drug abuser (current or previous)
* Psychiatric condition or language barriers
* Planned Intensive Care Recovery

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 540 (Actual)
Dates: Start 2018-08-15 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Shorter Length Of Hospitalization (LOH) | Up to 4 weeks after surgery
  Total amount of days spent in hospital

SECONDARY OUTCOMES:
Assessment of postoperative pain | At moment 24 hours after surgery
  Measurement of pain score post-operation will be obtained using clinical data gathered by the care team providing routine clinical care, and asking routine pain score questions. The scale used is the standard 1-10 pain scale, with 1 being no pain or very mild discomfort, and 10 being very severe pain.
Presence/Absence of nausea | At moment 0, 3, 6, 12 and 24 hours after surgery
  Treatment for postoperative nausea
Presence/Absence of vomiting | At moment 0, 3, 6, 12 and 24 hours after surgery
  Treatment for postoperative vomiting
Time to flatus | Up to 4 weeks after surgery
  Hours elapsed to event
Time to bowel movement | Up to 4 weeks after surgery
  Hours elapsed to event
Foley catheter removal | From 1 to 14days post surgery
  Time to Foley catheter removal postoperative
Time to drink | Up to 4 weeks after surgery
  Hours elapsed to event
Time to eating | Up to 4 weeks after surgery
  Hours elapsed to event
Time to walking | Up to 4 weeks after surgery
  Hours elapsed to event
Postoperative complications | Up to 2 weeks after surgery
  Rate measurement
Time to adjuvant treatment | 60 days
  Time participant receives adjuvant treatment, if needed (chemotherapy or radiation)
Readmission rates | Up to 21 days post surgery
  Readmissions to the hospital

CONTACTS AND LOCATIONS:
Overall Officials: Beihua Kong, MD.PhD., Principal Investigator — Qilu Hospital of Shandong University
Locations (1):
- Qilu Hospital of Shandong University, Jinan, Shandong, China

REFERENCES:
- [Derived] Xing N, Wang H, Huang Y, Peng J. Enhanced recovery after surgery program alleviates neutrophil-to-lymphocyte ratio and platelet-to-lymphocyte ratio in patients undergoing gynecological surgery. Front Med (Lausanne). 2023 Apr 17;10:1057923. doi: 10.3389/fmed.2023.1057923. eCollection 2023. PMID 37138751
- [Derived] Peng J, Dong R, Jiao J, Liu M, Zhang X, Bu H, Dong P, Zhao S, Xing N, Feng S, Yang X, Kong B. Enhanced Recovery After Surgery Impact on the Systemic Inflammatory Response of Patients Following Gynecological Oncology Surgery: A Prospective Randomized Study. Cancer Manag Res. 2021 Jun 1;13:4383-4392. doi: 10.2147/CMAR.S294718. eCollection 2021. PMID 34103993